CLINICAL TRIAL: NCT05581732
Title: Russian Prospective Open Comparative in Two Groups, Low-interventional Study on the Effect of the Oral Nutrition Supplement (ONS) "Nutrinidrink With Dietary Fiber" on the Health Indicators in Children With Cerebral Palsy (CP)
Brief Title: Study of the ONS "Nutrinidrink With Dietary Fiber" Use Effect on Some Health Indicators in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Enrollme.ru, LLC (Network)
Collaborators: Danone Nutricia (Industry)
Responsible Party: Sponsor
Other Study IDs: NOCP
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Nutrition; Quality of Life; Bioimpedance; Z-score
MeSH Terms: conditions — Cerebral Palsy | interventions — Dietary Fiber

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: 32 patients in the study group received supplemental nutritional support with ONS "Nutrinidrink with Dietary Fiber" in a pre-calculated amount daily throughout the study for 14-16 weeks. During the hospital stay, additional nutritional support was added to the patient's standard hospital diet (ATC table). On an outpatient basis, the patient received the required amount of ONS at his disposal and add it as a supplement to his/her usual and habitual diet between main meals.
  Interventions: Dietary Supplement: Nutrinidrink with Dietary Fiber
- Control: 24 patients in the control group adhered to the standard hospital diet (ATC table), and at discharge - the usual habitual diet

INTERVENTIONS:
Dietary Supplement: Nutrinidrink with Dietary Fiber — Nutrinidrink with Dietary Fiber is a specialized nutrition for children during illness and recovery period, as well as with increased protein and energy needs: mental and / or physical stress, chronic diseases, growth and / or weight deficiency
  Groups: Study

SUMMARY:
The goal of this low-interventional study was to study the effect of additional nutritional support with ONS "Nutrinidrink with dietary fiber" on the anthropometric parameters of patients and the dynamics of gastrointestinal symptoms in patients with cerebral palsy. Among the additional objectives were to study the quality of life, metabolic parameters and the dynamics of some functional parameters of patients. Possible adverse events were also studied and described.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cerebral palsy, spastic and hyperkinetic forms;
* Class of cerebral palsy GMFCS 2-3;
* Z-score BMI ≤ -1;
* The patient's ability to safely swallow liquid food;
* Availability of informed consent signed by the patient's legal representative for inclusion in the study and processing of personal data.

Exclusion Criteria:

* Individual intolerance to the investigational product components;
* Galactosemia;
* Allergy to cow's milk proteins and other food intolerances;
* Participation in another clinical study currently or in the past 30 days;
* Any other medical or non-medical reason that, in the physician's opinion, may prevent the patient from participating in the study.
* Deterioration of the patient's condition requiring his transfer to enteral or parenteral nutrition;
* Transfer of a patient to another hospital;
* Complications that could be caused by the investigational product (diarrhea, nausea, vomiting, allergies, etc.);
* Withdrawal for a safety reason
* Refusal of the patient (his legal representative) from further participation in the study and withdrawal of informed consent to participate in the study and the processing of personal data. At the same time, the exclusion of a patient from the study should not affect the nature of his therapy

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Boys and girls, aged 4-8 years with confirmed diagnosis of cerebral palsy, spastic and hyperkinetic forms (Class of cerebral palsy GMFCS 2-3) and Z-score BMI ≤ -1
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
BMI | during observation up to 16 weeks
  Body Mass Index
Z-score (BMI) | during observation up to 16 weeks
  Body mass index z-scores are measures of relative weight adjusted for child age and sex
Bioelectrical impedance analysis | during observation up to 16 weeks
  Device-based diagnostics to measure the voltage of weak electrical currents in order to calculate impedance (resistance) of the body
Gastrointestinal symptoms scale | during observation up to 16 weeks
  A patient reported 5 score questionnaire to evaluate frequency and severity of gastrointestinal symptoms with 1 - minimal symptom manifestation, 5 - maximal symptom manifestation
Martinet-Kushelevsky test | during observation up to 16 weeks
  Activity test to determine the level of physical abilities

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail A Getman, Dr, Study Director — Enrollme.ru
Locations (3):
- Russia (3):
  - Center for nutrition and biotechnology, Moscow
  - Scientific and Clinical Center for Children's Psychoneurology, Moscow
  - Child's Clinical Hospital by Ivanova, Samara